CLINICAL TRIAL: NCT05241483
Title: SETİNT AI-Diseases
Brief Title: Remote Patient Monitoring and Detection of Possible Diseases With Artificial Intelligence Telemedicine System
Acronym: AI - diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Setint AI Robotic Sistem Egitim ve Danısmanlık San. Tic. A.S. (Other Government)
Responsible Party: Principal Investigator, Sezgin SEZER, Artificial Intelligence Specialist, Setint AI Robotic Sistem Egitim ve Danısmanlık San. Tic. A.S.
Other Study IDs: SETİNT-AI-TURKEY
Record Dates: First submitted 2022-02-03; First posted 2022-02-15 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Predictive Value of Tests; Vital Signs; Laboratory Critical Values; Relative Value Scales; Reference Values
Keywords: test; laboratory; relative value; homecar; artificial intelligence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Biospecimen Retention: Samples Without DNA — fever, pulse, blood pressure, oxygen saturation, glucose measurement values
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- fever: Remote patient monitoring. fever values recorded by the patient in the system. Validation of pre-diagnosis results of AI systems to detect fever-related diseases.
  Interventions: Diagnostic Test: mesure valition
- pulse: Remote patient monitoring. pulse values recorded by the patient in the system. Validation of pre-diagnosis results of AI systems to detect fever-related diseases.
  Interventions: Diagnostic Test: mesure valition
- blood pressure: Remote patient monitoring. Blood pressure values recorded by the patient in the system. Validation of pre-diagnosis results of AI systems to detect fever-related diseases.
  Interventions: Diagnostic Test: mesure valition
- oxygen saturation: Remote patient monitoring. oxygen saturationvalues recorded by the patient in the system. Validation of pre-diagnosis results of AI systems to detect fever-related diseases.
  Interventions: Diagnostic Test: mesure valition
- glucose: Remote patient monitoring. glucose values recorded by the patient in the system. Validation of pre-diagnosis results of AI systems to detect fever-related diseases.
  Interventions: Diagnostic Test: mesure valition

INTERVENTIONS:
Diagnostic Test: mesure valition — Possible diseases that may occur as a result of the patient's vital values with artificial intelligence systems
  Other Names: doctor examination; patient complaints; patient symptoms; Vital values recorded by the patient in the system.

SUMMARY:
Remote patient monitoring and detection of possible diseases with Artificial Intelligence Telemedicine System

DETAILED DESCRIPTION:
Possible disease detection with artificial intelligence from the patient's vital values possible disease detection from the patient's examination records

ELIGIBILITY:
Inclusion Criteria:

* No Eligibility Criteria

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients registered in the SETINT AI artificial intelligence Telemedicine system
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-03-30 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Patient symptoms and disease confirmation | May - October 2021
  Her physician's patient symptom data were successfully matched to ICD-10 and other disease codes using the AI model.

CONTACTS AND LOCATIONS:
Overall Officials: Aykut COŞKUN, MD, Principal Investigator — SETINT AI Robotic Sistem Eğitim ve Danışmanlık San.Tic.A.Ş.; İsmail ÇELİK, MD, Principal Investigator — SETINT AI Robotic Sistem Eğitim ve Danışmanlık San.Tic.A.Ş.
Locations (1):
- Setint Ai, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided